CLINICAL TRIAL: NCT03036722
Title: Effect of Phytoestrogen-rich Flaxseeds on Decreasing Bone Turnover in Postmenopausal Women Aged Between 50 -70 Years.
Brief Title: Flaxseed Consumption and Bone Metabolism in Postmenopausal Women.
Acronym: FLAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Dr Daniel Commane, Principal Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UOReading
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Bone Loss, Age Realted; Post Menopausal
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flaxseed porridge group (Experimental): 22 volunteer will be given 80g of a pre prepared porridge meal containing 40 g of ground (flaxseed) to consume daily.
  Interventions: Other: Flaxseed
- Placebo control porridge group (Placebo Comparator): 22 volunteer will be given 78.5g preprepared control porridge matched for energy and fat content to consume daily ( Matching food products: 22g MCT (medium chain Triglyceride), 5.5g pure egg white powder, 11g cream of rice).
  Interventions: Other: Placebo control porridge

INTERVENTIONS:
Other: Flaxseed — Flaxseed is a member of the genus Linum in the family Linaceae. It is a food and fiber crop and it occurs in two basic varieties: brown and yellow or golden (also known as golden linseeds).
  Arms: Flaxseed porridge group
Other: Placebo control porridge — control porridge matched for energy and fat content.
  Arms: Placebo control porridge group

SUMMARY:
This proposed randomized double blinded, placebo-controlled, parallel trial; with two arms, in females aged 50-70 years, volunteers will be postmenopausal with a BMI between 25-35 kg/m2. This study aims to determine the benefits of phytoestrogen-rich flaxseeds on decreasing bone turnover in postmenopausal women aged over 50 years.

DETAILED DESCRIPTION:
Osteoporosis affects approximately 1 in 3 women over the age of 50 and accounts for more days spent in hospital than diabetes and breast cancer; amongst women of that age group. Aging, a sedentary lifestyle, a poor diet and smoking are all risk factors. A healthy diet (including food rich in calcium, vitamin D and phytoestrogens) may protect against osteoporosis and risk of fractures. Phytoestrogens in the diet are of putative benefit through and post the menopause. The term phytoestrogens describes a wide variety of plant food derived chemicals having a structure similar to estradiol (oestrogen). The three main classes of phytoestrogens are the isoflavones, the lignans and coumestans. Oil seeds are a good source of lignans, with flaxseeds being particularly rich. Flaxseeds consumption has previously been associated with changes in bone turnover markers in postmenopausal women.

This study therefore is designed to test the hypothesis that consumption of a quantity of flaxseeds achievable in an individual's habitual diet (40g) will induce improvements in bone turnover markers, mediated through the increased circulation of phytoestrogens, in postmenopausal women.

. The study arms are i) A placebo control arm, volunteers consume a placebo 40g porridge (matched for fibre and fat with the flaxseed product) every day over 12 weeks, or ii) 40g of flaxseeds added to 40g porridge daily over a 12 week study period. Adherence to the intervention will be assessed via analysis of concentrations of the mammalian lignans enterolactone and enterodiol in urine. The primary outcome for the study will be changes in markers of bone health. The secondary outcomes for the study will be changes in urinary and plasma androgens. Volunteers will need to attend the Hugh Sinclair Unit of Human Nutrition clinical unit on four occasions to facilitate screening and the study visit.

Volunteers will be required to provide a fasting blood (30ml; 2 tablespoons); 24 hr urine (started the day prior to each study visit) and faecal samples at all 3 study visits (baseline, weeks 6 and 12). As vitamin D status and bone turnover markers are related to bone health, the volunteers will be given the opportunity to undergo an additional measurement of total body composition using dual-energy x-ray absorptiometry (DXA) at baseline and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (self reported of final menstrual cycle occurred at least 1 year ago).
* 50-70 years.
* BMI ≥25-35 kg/m2.
* Fasting serum Glucose <7 mmol/l (not diagnosed with diabetes)
* Fasting total cholesterol<7.8 mmol/l and triacylglycerol <2.3 mmol/l.
* Normal liver and kidney function (assessed by measuring total bilirubin, uric acid, creatinine and liver enzymes in the screening blood sample).
* Not having suffered fractures of the hip, wrist or spine, osteoporosis or osteomalacia.
* Blood pressure lower than BP <140/90 mmHg.
* Not having any medical related cause that influencing bone turnover; these include:

  * Steroid medical treatment, e.g. 5 mg/ day of prednisolone.
  * Abnormal hormonal fluctuation women who self-reported previous diagnoses of thyroid disease, Thyroid hormonal abnormalities, progesterone and oestrogen high level.
  * Diagnosed with vitamin D deficiency.
* Not suffering any cardiovascular diseases/ heart diseases e.g. stroke in the past 12 months.
* Not using hormone replacement medicine e.g. oestrogen.
* Not using any calcium or vitamin D supplements during the last 3 months.
* Not suffering from renal or bowel disease.
* No history of alcohol misuse based on self-reported alcohol intake and measurement of liver enzymes in the screening blood sample.

Exclusion Criteria:

* Women who became menopausal as the result of surgery (e.x. removal of both ovaries).
* Current smoker.
* Anaemic, haemoglobin ≤ 115g/l or who have abnormal blood biochemistry based on standard clinical cut- offs.
* Have history of food intolerances/allergies (e.g. gluten or dairy) or intolerances (e.g. lactose).
* Received antibiotics in the previous six months.
* Trying to lose weight by following a diet or exercise regimen designed for weight loss, or taking any drug influencing appetite and any drug for weight loss for the last three months.
* Have participated in similar dietary or probiotics-containing product's clinical trials within 3 months before the screening visit.
* Using soy/isoflavone, flax oil and flax supplements.
* Using prebiotic / probiotic during the last 6 months.
* Excessive exercise more than three times a week, including weight bearing exercise.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Determine the benefits of phytoestrogen-rich flaxseeds on decreasing bone turnover in postmenopausal women. | 12 weeks
  To observe the effect of consuming 40g of flaxseeds/ daily for 12 weeks on bone health of postmenopausal women by measuring some markers of bone resorption and formation 3 during the study period (baseline, 6 and 12 week)

SECONDARY OUTCOMES:
Gut microbial | 12 weeks
  Observe the role of gut microbial on flaxseed metabolite.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Proven, PhD, Study Chair — Ethics committee Co-ordinator
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cosman F, de Beur SJ, LeBoff MS, Lewiecki EM, Tanner B, Randall S, Lindsay R; National Osteoporosis Foundation. Clinician's Guide to Prevention and Treatment of Osteoporosis. Osteoporos Int. 2014 Oct;25(10):2359-81. doi: 10.1007/s00198-014-2794-2. Epub 2014 Aug 15. PMID 25182228
- [Background] Foundation, N. O. (2003). Physician's guide to prevention and treatment of osteoporosis, National Osteoporosis Foundation.
- [Background] Hutchins AM, Martini MC, Olson BA, Thomas W, Slavin JL. Flaxseed consumption influences endogenous hormone concentrations in postmenopausal women. Nutr Cancer. 2001;39(1):58-65. doi: 10.1207/S15327914nc391_8. PMID 11588903
- [Background] Mei J, Yeung SS, Kung AW. High dietary phytoestrogen intake is associated with higher bone mineral density in postmenopausal but not premenopausal women. J Clin Endocrinol Metab. 2001 Nov;86(11):5217-21. doi: 10.1210/jcem.86.11.8040. PMID 11701680
- [Background] Weaver CM, Cheong JM. Soy isoflavones and bone health: the relationship is still unclear. J Nutr. 2005 May;135(5):1243-7. doi: 10.1093/jn/135.5.1243. PMID 15867312
- [Background] Go G, Tserendejid Z, Lim Y, Jung S, Min Y, Park H. The association of dietary quality and food group intake patterns with bone health status among Korean postmenopausal women: a study using the 2010 Korean National Health and Nutrition Examination Survey Data. Nutr Res Pract. 2014 Dec;8(6):662-9. doi: 10.4162/nrp.2014.8.6.662. Epub 2014 Sep 15. PMID 25489406